CLINICAL TRIAL: NCT01004159
Title: A Phase II Study of High Dose Cetuximab Plus Irinotecan in Colorectal Cancer Patients With KRS-Wild Type Tumors Who Progressed After Failure of Prior Standard Dose ofCetuximab Plus Irinotecan
Brief Title: Cetuximab Plus Irinotecan in Colorectal Cancer Patients Who Progressed After Failure With Cetuximab Plus Irinotecan
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: former PI left institute
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 152009
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; KRAS wild type tumors
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cetuximab with irinotecan (Experimental)
  Interventions: Drug: cetuximab with irinotecan

INTERVENTIONS:
Drug: cetuximab with irinotecan — Cetuximab administered 500mg/m2 over 120 minutes Irinotecan administered Q 3 weeks, Q 2 weeks or Q week x 4 every 6 weeks depending on patients previous treatment

SUMMARY:
This study is being performed to test if the use of high dose of cetuximab in combination with irinotecan overcomes the resistance seen with standard dose of cetuximab plus irinotecan in patients with wild type KRS tumors that have advanced colon or rectal cancer

DETAILED DESCRIPTION:
Cetuximab is a manufactured antibody-antibodies are proteins that can be found circulating in your blood stream. The growth of colorectal cancer may be affected by the interaction of a growth factor known as "epidermal growth factor" (EGF) with its receptor.

Cetuximab is a antibody directed against the receptor for EGF and has been shown to turn off the activity of the receptor and to stop the growth of cancer cells in many laboratory tests. Cetuximab has been recently approved by the Food and Drug Administration in the treatment of patients with advanced colorectal cancer and who failed standard chemotherapy. Cetuximab has been shown to delay the progression of colorectal cancer when given alone in patients who have failed standard chemotherapy and when given with a chemotherapy drug called irinotecan in patients who have failed irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colon cancer that is metastatic or unresectable
* Progressed on cetuximab plus irinotecan based combination prior to enrolling on this study
* Patient must have tumor tissue tested for KRAS mutation and should be confirmed to carry a wild type
* ECOG less than or equal to 1
* Must have adequate organ and marrow function
* Ability to understand and the willingness to sign a written informed consent document.
* Presence of measurable disease defined as a lesion ≥ 2 cm by CT (or 1 cm by spiral CT). All sites of disease should be evaluated ≤ 3 weeks before treatment initiation
* Patients should have failed or been deemed intolerant to other standard chemotherapy treatments such as oxaliplatin and fluoropyrimidines

Exclusion Criteria:

* Patients may not be receiving any other investigational agents that are not included in this study. Prior investigational anticancer agents wil not be allowed within 4 weeks prior to study treatment. Herbal medicine and vitamins wil not be considered as contraindications for enrollment on study.
* Patients with known brain metastases are not eligible unless brain metastases are treated and stable on radiographic follow-up and without significant symptomatology
* History of other invasive cancers with current evidence of disease
* Patients should be off chemotherapy or other targeted therapies for at least 3 weeks before study treatment. Mitomycin C treatment should be at least 6 weeks before study treatment
* History of allergic reactions to irinotecan
* Prior severe infusion reaction to cetuximab
* History of allergic reaction to tetracycline or doxycycline
* Need for prior dose reduction on cetuximab secondary to grade 3 skin toxicity
* Active skin toxicity of grade 2 or higher at the time of study enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the chemotherapeutic agents proposed are category D agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued if the mother is treated on this study.
* Grade 2 or higher hypomagnesemia at baseline evaluation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: WenWee Ma, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab With Irinotecan
Started | 20
Completed | 0
Not Completed | 20
Not completed — Adverse Event | 2
Not completed — Disease Progression | 18

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Cetuximab With Irinotecan
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (10.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: 12-week Progression Free Survival Rate Upon Escalation of Cetuximab Dose to 500mg/m2 in Combination With Irinotecan After Progression on Standard Dose Therapy in Patients With KRS Wild Type Colorectal Cancer
Time Frame: 12 week
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab With Irinotecan
Number analyzed (Participants) | 20
percentage of participants | 50 [27 to 69]

2. Secondary Outcome: Response Rate of Cetuximab 500mg/m2/Week in Combination With Irinotecan in the Enrolled Patient Population
Time Frame: 18 months
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of particitpants
Arm/Group | Cetuximab With Irinotecan
Number analyzed (Participants) | 20
percentage of particitpants | 5 [.1 to 24.9]

ADVERSE EVENTS:
Arm/Group | Cetuximab With Irinotecan
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab With Irinotecan (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Pain (General disorders) | 1 (2)
Hypersensitivity (Immune system disorders) | 1 (2)
Infection (Infections and infestations) | 2 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab With Irinotecan (N=20)
Leukopenia (Blood and lymphatic system disorders) | 4 (12)
Lymphopenia (Blood and lymphatic system disorders) | 4 (24)
Neutropenia (Blood and lymphatic system disorders) | 3 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Dry eye (Eye disorders) | 1 (2)
Lacrimation increased (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (10)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (6)
Oral pain (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (8)
Fatigue (General disorders) | 3 (8)
Mucosal inflammation (General disorders) | 1 (2)
Pyrexia (General disorders) | 1 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (6)
Herpes zoster (Infections and infestations) | 1 (2)
Infection (Infections and infestations) | 2 (6)
Laceration (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (6)
Blood alkaline phosphatase increased (Investigations) | 3 (8)
Blood bilirubin increased (Investigations) | 1 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (2)
Haemoglobin (Investigations) | 1 (6)
Haemoglobin decreased (Investigations) | 2 (16)
International normalised ratio (Investigations) | 1 (2)
International normalised ratio increased (Investigations) | 1 (4)
Weight decreased (Investigations) | 3 (6)
Anorexia (Metabolism and nutrition disorders) | 6 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (16)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (58)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (4)
Restless legs syndrome (Nervous system disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (4)
Mood altered (Psychiatric disorders) | 1 (2)
Bladder pain (Renal and urinary disorders) | 1 (2)
Haematospermia (Reproductive system and breast disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (4)
Hypotension (Vascular disorders) | 2 (4)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes